CLINICAL TRIAL: NCT06742866
Title: The Efficacy and Safety of Intravenous + Oral Vs. Oral Amiodarone in Preventing Recurrence After Catheter Ablation in Patients with Persistent Atrial Fibrillation
Brief Title: Efficacy and Safety of Intravenous + Oral Vs. Oral Amiodarone in Preventing Recurrence After Catheter Ablation in Patients with Persistent Atrial Fibrillation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITAD-PAF
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Intravenous + Oral Amiodarone) (Experimental): Within 24 hours post-operation, patients will receive an intravenous amiodarone loading dose of 300 mg QD along with oral amiodarone 200 mg BID. This regimen will be continued for 3 days, after which intravenous amiodarone will be discontinued, and oral amiodarone 200 mg BID will be continued for 3 months.
  Interventions: Drug: Amiodarone Injection
- Control group (Oral Amiodarone only) (Placebo Comparator): Postoperatively, instead of administering intravenous amiodarone, sodium chloride injection was used as a placebo, and oral amiodarone 200 mg BID was directly given for 3 months.
  Interventions: Drug: Sodium Chloride Injection 0.9%

INTERVENTIONS:
Drug: Amiodarone Injection — Administer 300 mg of intravenous amiodarone as a loading dose once daily (QD) and 200 mg of oral amiodarone twice daily (BID) within 24 hours postoperatively, and continue for 3 consecutive days.
  Arms: Experimental group (Intravenous + Oral Amiodarone)
Drug: Sodium Chloride Injection 0.9% — Sodium chloride injection as a placebo in an amount equivalent to amiodarone injection.
  Arms: Control group (Oral Amiodarone only)

SUMMARY:
This study aims to investigate the efficacy and safety of intravenous combined with oral amiodarone in preventing atrial fibrillation (AF) recurrence after catheter ablation in patients with persistent atrial fibrillation. Using a randomized controlled trial design, patients will be divided into two groups: intravenous + oral amiodarone and oral amiodarone alone. Through multiple follow-ups at 1, 3, 6, and 12 months post-procedure, the study will compare the two treatment regimens in terms of blood concentrations of amiodarone and its metabolites, efficacy (short-term recurrence [SR], long-term recurrence [LR], and patient quality of life), and safety (adverse drug reactions). Subgroup analyses will also be conducted to explore potential differences in drug treatment effects among populations with varying risk factors. This study aims to provide valuable clinical data for post-ablation management of atrial fibrillation, contributing to the development of optimized treatment strategies to enhance therapeutic outcomes and improve patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥18 years;
* First-time catheter ablation for persistent atrial fibrillation (defined as any - previous episode lasting ≥7 days);
* Symptomatic atrial fibrillation patients who have failed or are intolerant to at least one class I or III antiarrhythmic drug;
* Participants who are able to understand the purpose of the study, voluntarily agree to participate, and provide written informed consent.

Exclusion Criteria:

* Those unwilling or unsuitable to restart or continue antiarrhythmic drug therapy;
* Life expectancy < 12 months;
* Severe liver or kidney dysfunction;
* Allergy to amiodarone components;
* Pregnant or breastfeeding women;
* Contraindications to amiodarone (e.g., blood pressure < 90/60 mmHg; bradycardia < 55 bpm, second- or third-degree AV block, or sick sinus syndrome);
* Thyroid disorders, such as hyperthyroidism or hypothyroidism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2024-12-16 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial arrhythmia lasting more than 30 seconds. | At least 12 months of follow-up, beyond the initial 3 month blanking period
  After a single ablation procedure, with at least 12 months of follow-up, any atrial arrhythmia recorded for more than 30 seconds - including atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL) - occurring beyond the initial 3-month blanking period.

SECONDARY OUTCOMES:
Recurrence of atrial fibrillation (AF) lasting more than 30 seconds. | At least 12 months of follow-up, beyond the initial 3 month blanking period
  After a single ablation procedure, with at least 12 months of follow-up, any atrial arrhythmia recorded for more than 30 seconds - including atrial fibrillation (AF) - occurring beyond the initial 3-month blanking period.
Recurrence of atrial arrhythmias during the 3-month blanking period after atrial fibrillation (AF) surgery. | During the 3-month blanking period after atrial fibrillation (AF) surgery
  Recurrence of atrial arrhythmias during the 3-month blanking period after atrial fibrillation (AF) surgery.
hospital readmission for re-ablation, electrical cardioversion and adverse drug events (ADEs) | At least 12 months of follow-up
  During the follow-up period, hospital readmission for re-ablation, electrical cardioversion and adverse drug events (ADEs), including bleeding, liver dysfunction, renal dysfunction, skin sensitivity, gastrointestinal adverse reactions, bradyarrhythmia (<55 bpm), ischemic stroke, and hyperthyroidism, etc.
Quality of life assessment using AFEQT | At least 12 months of follow-up
  Assessment of quality of life using the AFEQT (Atrial Fibrillation Effect on Quality of Life Questionnaire) during at least 12 months of follow-up.
Serum drug concentrations of amiodarone and its metabolite desethylamiodarone. | At 1 month and 3 months after surgery.
  Serum drug concentrations of amiodarone and its metabolite desethylamiodarone at 1 month and 3 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Xuhui, China